CLINICAL TRIAL: NCT03116789
Title: Analysis of Ameliorative Effects of Oral Probiotics on Bacterial Vaginosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GenMont Biotech Incorporation (Industry)
Collaborators: Kuo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NP105004
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Randomized, Parallel, open lable Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VGA-1(Probiotics) (Active Comparator): Lactobacillus rhamnosus and Lactobacillus acidophilus.
  Interventions: Dietary Supplement: probiotics
- VGA-2(Probiotics) (Active Comparator): Lactobacillus rhamnosus and Lactobacillus plantarum.
  Interventions: Dietary Supplement: probiotics

INTERVENTIONS:
Dietary Supplement: probiotics — Two capsules for daily

SUMMARY:
The purpose of this study is to analyze the ameliorative effects of oral probiotics on bacterial vaginosis.

DETAILED DESCRIPTION:
To analyze the oral Lactobacillus rhamnosus with Lactobacillus acidophilus or Lactobacillus rhamnosus with Lactobacillus plantarum could be ameliorative effects for bacterial vaginosis.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent Form.
* Subjects with bacterial vaginosis and Nugent score as 4-10
* Subjects in age of 20-55 years old
* Regularly menstruating premenopausal women (normal menstrual function (Eumenorrhoea) shall mean regular menstrual bleeding pattern every 28 plus/minus 10 days)
* Forbidden sexual behavior was required 72 hours before all visits

Exclusion Criteria:

* Subjects are pregnant, lactating or planning to become pregnant.
* Allergy to test products (raw material components included: Anhydrous glucose, Magnesium stearate, Fructooligosaccharides, Microcrystalline cellulose, Lactobacillus, etc.)
* Bleeding from genital tract of unknown aetiology.
* Congenital and acquired immunodeficiencies.
* Diabetes
* Mental illness
* Malignant tumor
* Application of NuvaRing hormonal contraceptive vaginal ring
* Application of mechanical contraceptives, such as: diaphragms, intrauterine contraceptive insert, except condom
* Application of hormonal preparations, such as: Vagifem, Ovestin and vaginal estrogens in reproductive period.
* Mycotic vaginitis
* Antibiotic(unless indicated by PI) and steroids therapy during this trial.
* Use of oral or vaginal probiotic products (sachet, capsule, or tablet) four weeks before V1.
* Participation in another clinical study.

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Nugent Score | 4 weeks
  The degree of decline for Nugent score

SECONDARY OUTCOMES:
Vaginal pH | 4 weeks
  Vaginal pH value changes
Vaginal secretions microflora | 4 weeks
  Changes in vaginal secretions microflora

CONTACTS AND LOCATIONS:
Overall Officials: Ta-Chin Lin, Principal Investigator — Kuo General Hospital
Locations (1):
- KUO general hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided